CLINICAL TRIAL: NCT02492477
Title: TOP-TRIAL The Safety of Not Flushing the Non-used PORT-A-CATH® in Cancer Patients - a Prospective, Two-arm Phase I Trial, Pilot Trial
Brief Title: TOP-TRIAL Safety of Not Flushing Non-used PORT-A-CATH® in Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Krankenhaus Barmherzige Schwestern Linz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TOP-TRIAL-2014-1.2
Record Dates: First submitted 2015-06-29; First posted 2015-07-08 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Adjuvant Chemotherapy; Solid Tumours; Port-A-Cath
MeSH Terms: interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6 months (Experimental): evaluation of PORT-A-CATH®, blocking with Medunasal®-Heparinblock, restoration of PORT-A-CATH® with Alteplase
  Interventions: Procedure: evaluation of PORT-A-CATH®; Drug: blocking with Medunasal®-Heparinblock; Drug: restoration of PORT-A-CATH® with Alteplase
- 12 months (Experimental): evaluation of PORT-A-CATH®, blocking with Medunasal®-Heparinblock, restoration of PORT-A-CATH® with Alteplase
  Interventions: Procedure: evaluation of PORT-A-CATH®; Drug: blocking with Medunasal®-Heparinblock; Drug: restoration of PORT-A-CATH® with Alteplase

INTERVENTIONS:
Procedure: evaluation of PORT-A-CATH® — in patients in curative setting, clinical assessment, PORT-A-CATH® testing of possibility of saline-administration and blood withdrawal with vacutainer, laboratory assessment
Drug: blocking with Medunasal®-Heparinblock — blocking of the functioning PORT-A-CATH® with heparinized 0,9% NaCl solution
  Other Names: heparinized 0,9% NaCl solution
Drug: restoration of PORT-A-CATH® with Alteplase — by malfunction of the PORT-A-CATH® attempting of restoration with Actilyse® according to guidelines
  Other Names: Actilyse®

SUMMARY:
The benefits and risks of flushing or not flushing the non-used PORT-A-CATH® in cancer patients and the time interval of eventual PORT-A-CATH® flushing are currently unknown. The manufacturers of PORT-A-CATH® recommend regular flushings every 4 weeks. In clinical practice, the intervals are usually at least three months. Regular flushing might lead to a decreased risk of PORT-A-CATH® thrombosis, but may also lead to an increased infection or thrombosis rate and patients discomfort. Therefore, this study investigates the safety of not flushing the PORT-A-CATH® for 6 or 12 months.

DETAILED DESCRIPTION:
Currently it is unknown if flushing a non-used PORT-A-CATH® every 4 weeks is a valid strategy to preserve its functioning. Even more, decision to keep the PORT-A-CATH® after completion of adjuvant therapy cannot be based on profound patient information as there exist hardly any data regarding PORT-A-CATH® related complications of non-used PORT-A-CATH®.

The proposed prospective, two arm trial aims to investigate if no flushing of a non-used PORT-A-CATH® over a period of one year has equal PORT-A-CATH® related complications compared to flushing the PORT-A-CATH® every 4 weeks.

The proposed trial also aims to examine the frequencies of PORT-A-CATH® related complications in non-used PORT-A-CATH®. The authors put up the hypothesis that there will be fewer port-a-cath related infections in the experimental arms compared to the infection rate mentioned in the literature up to 27 %, since the puncture of the PORT-A-CATH® and the administration of fluids are the main causes of infection.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients in curative setting, with port a cath Implantation for systemic chemotherapy, including neo-adjuvant and adjuvant chemo-immunotherapy and supportive therapy (e.g. parenteral Nutrition)
* Completion of curative Treatment with port a cath indication, operation included, regardless of a non-intravenous (subcutaneous or oral) given therapy (endocrine therapy, chemo-immunotherapy, radiotherapy)
* patients with pectoral port a cath systems
* No port a cath associated complications during curative therapy such as investigated events: persistent malfunction, thrombosis, infection of the port-a-cath (to puncture the port a cath under X-ray control is allowed except it results in diangosis of persistent malfunction)
* No therapeutic anticoagulant therapy (phenprocoumon/Marcoumar®, heparin)
* No evidence of metastatic disease
* ≥18 years
* Willing to participate

Exclusion Criteria:

* No signed informed consent
* Patients with port a cath systems other than pectoral port a cath systems (e.g. forearm port a cath System)
* Unable to attend control timepoints
* Use of the port-a-cath after the above defined curative treatment (within the investigational period)
* Willing to explant the port-a-cath
* Willing to become pregnant within one year after adjuvant treatment
* Patient with heparin-induced Thrombocytopenia (HIT)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
incidences of PORT-A-CATH® related events (persistent malfunction, thrombosis, infection) | 6 or 12 months

SECONDARY OUTCOMES:
incidences of restoration of PORT-A-CATH® function by alteplase | 6 or 12 months
rate of necessary PORT-A-CATH® removal | 6 or 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Judith Lafleur, OA Dr., Principal Investigator — BHSL, Abt. für Gynäkologie
Locations (1):
- Krankenhaus der Barmherzigen Schwerstern Linz Betriebsges.m.b.H., Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No